CLINICAL TRIAL: NCT07175480
Title: An Open-label, Investigator-initiated, Single Arm, Exploratory Phase 2 Trial Evaluating the Feasibility and Efficiency of PET/CT Directed Free of Therapy Used for Metastatic and Advanced Renal Cell Carcinoma
Brief Title: PET/CT-Directed Free of Therapy for Metastatic RCC Patients With IMDC Favorable or Intermediate Risk
Acronym: Perfumer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025DZKY-069-01
Record Dates: First submitted 2025-08-30; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma (RCC); Metastatic Renal Cell Carcinoma (mRCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment pause (Experimental): Patients achieving complete metabolic response (CMR) or partial metabolic response (PMR) on PET/CT within 24 months discontinue combination regimens with the possibility to restart initial treatment at progression.
  Interventions: Drug: Intermittent PD-1/PD-L1 ICI + VEGFR-TKI

INTERVENTIONS:
Drug: Intermittent PD-1/PD-L1 ICI + VEGFR-TKI — Any PD-1/PD-L1 inhibitor or VEGFR-TKI that is commercially marketed, regulatory-approved and reimbursed under public health plans.Dose as recommended by the manufacturer.
  Other Names: Treatment pause

SUMMARY:
This phase 2 trial aims to test the feasibility and efficiency of PET/CT-directed treatment interruption strategy in metastatic renal cell carcinoma patients with IMDC favorable/intermediate risk who achieve complete (CMR) or partial metabolic response (PMR) after ≥12 months of first-line PD-1/PD-L1 Immune checkpoint inhibitor (ICI)+ VEGFR-tyrosine kinase inhibitor (TKI) therapy. It helps figure out whether PET/CT can safely direct treatment pause as well as explores a new individualized treatment option based on metabolic imaging for RCC patients.

DETAILED DESCRIPTION:
Current first-line therapy for advanced renal cell carcinoma (RCC) combines tyrosine kinase inhibitors (TKIs) with immune checkpoint inhibitors (ICIs). Although effective, continuous treatment often results in cumulative toxicities, significant financial burdens, and potential overtreatment for patients.

To improve such limitations, intermittent therapy strategies has gained more attention. However, existing approaches are constrained by insufficient induction periods (<12 months) that may compromise treatment depth, and reliance on anatomic CT criteria (RECIST 1.1) which cannot reliably differentiate residual active tumor from treatment-related fibrosis/necrosis. PET/CT quantifies tumor metabolic activity via standardized uptake values (SUV), enabling early molecular-level response assessment per PERCIST 1.0 criteria, thus shows promising prospects.

This trial implements a two-stage screening approach. During the pre-screening period, eligible unresectable/metastatic RCC patients with IMDC low/intermediate risk sign the Pre-screening Consent Form to receive ≥12 months of standard ICI+TKI therapy. Consolidative surgery and consolidative radiotherapy during combination therapy are permitted. Patients achieving complete metabolic response (CMR) or partial metabolic response (PMR) on PET/CT within 24 months undergo main screening. Those qualifying sign the Informed Consent Form (ICF), discontinue both agents and enter a closely monitored treatment holiday. During this phase, serial imaging (CT with supplemental PET/CT when indicated) will be performed every 12 ± 1 weeks. Therapy will be restarted immediately if any of the following occur:

* A ≥10% increase in the sum of the longest diameters (SLD) of target lesions from nadir, concurrent with a ≥30% increase in the peak standardized uptake value normalized to lean body mass (SULpeak) relative to baseline;
* New lesion with SULpeak exceeding liver background.

Peripheral blood and other biological samples from participants at different time points during the trial will be collected for future analyses. The primary endpoint is progression-free survival (PFS) rate at 24 months from treatment initiation. Secondary endpoints include duration of response after interruption, objective response rate after restarting therapy, safety (CTCAE v5.0-graded adverse events), patient-reported outcomes and cost-effectiveness. This study pioneers metabolic imaging to guide intermittent therapy in mRCC patients, utilizing extended induction and dual anatomic/metabolic restart thresholds to optimize risk-benefit balance while reducing treatment burden.

ELIGIBILITY:
Pre-screening Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years at time of signing informed consent
2. Locally advanced (not amenable to curative surgery or radiation therapy) or metastatic RCC (American Joint Committee on Cancer [AJCC] Stage IV)
3. Favorable or intermediate risk as per International Metastatic RCC Database Consortium (IMDC) criteria
4. Eastern Cooperative Oncology Group performance status 0 or 1
5. Karnofsky Performance Status (KPS) grade ≥ 70%
6. Adequate organ and bone marrow function meeting all laboratory criteria:

   Ⅰ. Absolute neutrophil count (ANC) ≥ 1.5 × 10³/μL (≥ 1.5 GI/L); Platelet count ≥ 100 × 10³/μL (≥ 100 GI/L); Hemoglobin ≥ 9 g/dL (≥ 90 g/L)

   Ⅱ. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × upper limit of normal. Total bilirubin ≤ 1.5 × the upper limit of normal (≤ 3 mg/dL [≤ 51.3 μmol/L] if Gilbert's syndrome)

   Ⅲ. Serum creatinine ≤ 2.0 × upper limit of normal or calculated creatinine clearance ≥ 30 mL/min using the Cockroft-Gault formula.
7. Capacity to comprehend and comply with protocol requirements, with documented informed consent signed
8. Contraception agreement for sexually active fertile participants and partners to use of medically accepted methods during study and continue for 5 months after last treatment
9. Negative pregnancy status at screening for women of childbearing potential

Pre-screening Exclusion Criteria:

1. Highly malignant pathology
2. Prior systemic therapy for advanced RCC
3. Poor risk as per International Metastatic RCC Database Consortium (IMDC) criteria
4. ECOG performance status >1
5. Karnofsky Performance Status (KPS) <70%
6. Inadequate organ and bone marrow function
7. Bulky or symptomatic disease or hepatic metastases
8. Active brain metastases or leptomeningeal disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before the start of treatment.
9. Concurrent or prior invasive malignancies that could confound efficacy assessment, except adequately treated non-melanoma skin cancer, superficial bladder cancer or carcinoma in situ of the cervix/breast with curative therapy >3 years ago.
10. Uncontrolled hypertension (>150/100 mmHg despite optimal therapy)
11. Uncontrolled comorbidities within 6 months including but not limited to: clinically significant cardiovascular disorders, gastrointestinal disorders with high risk of perforation or fistula formation, significant hematuria, hematemesis, hemoptysis, or major bleeding history, severe infections, severe autoimmune diseases (e.g., systemic lupus erythematosus, immune pneumonitis), active HIV, HBV, or HCV infections.
12. Major surgery within 4 weeks with unhealed wounds or planned surgery during study
13. Concomitant use of drugs or substances affecting activity or pharmacokinetics of investigational products
14. Hypersensitivity to any component of study drugs
15. Chronic or concurrent immunosuppressive therapy, except Inhaled/topical steroids
16. Medical/psychiatric/social conditions compromising protocol compliance
17. Pregnancy, lactation, or refusal of contraception during and for 5 months post-treatment
18. Inability to undergo PET/CT or oral drug administration

Main-screening Inclusion Criteria:

1. Patient must receive≥12 months of first line treatment with the combination of PD-1/PD-L1 ICI and VEGFR-TKI, and have not experienced a toxicity that prevents them from continuing on therapy.
2. Patients must achieve complete metabolic response (CMR) or partial metabolic response (PMR) on PET/CT within 24 months of the combination treatment with PD-1/PD-L1 ICI and VEGFR-TKI.
3. Favorable or intermediate risk as per International Metastatic RCC Database Consortium (IMDC) criteria
4. Eastern Cooperative Oncology Group performance status 0 or 1
5. Karnofsky Performance Status (KPS) grade ≥ 70%
6. Adequate organ and bone marrow function meeting all laboratory criteria:

   Ⅰ. Absolute neutrophil count (ANC) ≥ 1.5 × 10³/μL (≥ 1.5 GI/L); Platelet count ≥ 100 × 10³/μL (≥ 100 GI/L); Hemoglobin ≥ 9 g/dL (≥ 90 g/L)

   Ⅱ. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × upper limit of normal. Total bilirubin ≤ 1.5 × the upper limit of normal (≤ 3 mg/dL [≤ 51.3 μmol/L] if Gilbert's syndrome)

   Ⅲ. Serum creatinine ≤ 2.0 × upper limit of normal or calculated creatinine clearance ≥ 30 mL/min using the Cockroft-Gault formula.
7. Capacity to comprehend and comply with protocol requirements, with documented informed consent signed
8. Contraception agreement for sexually active fertile participants and partners to use of medically accepted methods during study and continue for 5 months after last treatment
9. Negative pregnancy status at screening for women of childbearing potential

Main-screening Exclusion Criteria:

1. Failure to complete ≥12 months of first-line PD-1/PD-L1 + VEGFR-TKI therapy due to unmanageable toxicity or other reasons
2. Failure to achieve CMR or PMR on PET/CT within 24 months after combination therapy; new metastatic lesions or disease progression on PET/CT.
3. Poor risk as per International Metastatic RCC Database Consortium (IMDC) criteria
4. ECOG performance status >1
5. Karnofsky Performance Status (KPS) <70%
6. Inadequate organ and bone marrow function
7. Uncontrolled hypertension (>150/100 mmHg despite optimal therapy)
8. Uncontrolled comorbidities including but not limited to: clinically significant cardiovascular disorders, gastrointestinal disorders with high risk of perforation or fistula formation, significant hematuria, hematemesis, hemoptysis, or major bleeding history, severe infections, severe autoimmune diseases (e.g., systemic lupus erythematosus, immune pneumonitis), active HIV, HBV, or HCV infections.
9. Medical/psychiatric/social conditions compromising protocol compliance
10. Pregnancy, lactation, or refusal of contraception during study period.
11. Inability to undergo PET/CT or oral drug administration

Withdrawal Criteria:

1. Disease progression with unsatisfactory efficacy, or occurrence of intercurrent illnesses during treatment or follow-up period.
2. Occurrence of severe treatment-related adverse reactions.
3. Laboratory test results indicating critical safety values.
4. Voluntary withdrawal of informed consent by the patient.
5. Investigator's judgment that withdrawal is in the subject's best interest.
6. Pregnancy during the trial period.
7. Wrong Enrollees: deviation of inclusion or exclusion criteria.
8. Poor patient compliance.
9. Loss to follow-up or death during the trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | 24 months from treatment initiation
  Proportion of participants alive and without disease progression at 24 months will be assessed according to PERCIST 1.0 criteria.

SECONDARY OUTCOMES:
Duration of response (DoR) | From treatment interruption until disease progression or death, assessed up to 24 months
  Time from first documented complete metabolic response (CMR) or partial metabolic response (PMR) to disease progression or death.
Overall survival (OS) | From treatment initiation until death from any cause, assessed up to 5 years
  Time from date of enrollment to date of death due to any cause.
Progression free survival (PFS) | From treatment initiation until disease progression or death from any cause, assessed up to 5 years
  Time from first study drug administration to first documented objective disease progression (PD) or death, whichever occurs first.
Overall safety profile | From the date of the first study drugs administration up to 90 days after the last dose of study drugs administration
  Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 criteria.
Patient-reported outcome (PRO) - Health-related quality of life measured by NCCN FKSI-19 | 24 months from treatment initiation
  Measured by the NCCN functional assessment of cancer therapy-kidney symptom index (FKSI-19), a 19-item scale assessing treatment-related symptoms and side effects for kidney cancer patients.
Patient-reported outcome (PRO) - Health-related quality of life measured by EORTC QLQ-C30 | 24 months from treatment initiation
  Measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30), a 30-item instrument assessing various domains of physical, emotional, and social functioning for cancer patients.
Patient-reported outcome (PRO) - General Health status measured by EQ-5D-5L | 24 months from treatment initiation
  Measured by the "5-Level EuroQol Group's 5-Dimension" (EQ-5D-5L) questionnaire which comprises the EQ-5D index evaluating health across five dimensions and the EQ-VAS which is a 0-100 visual scale for self-rated overall health.
Patient-reported outcome (PRO) - Anxiety and depression status measured by HADS | 24 months from treatment initiation
  Measured by the Hospital Anxiety and Depression Scale (HADS) which contains 14 items with 7 items measuring anxiety level and 7 items measuring depression level.
Quality-adjusted life years (QALYs) | 24 months from treatment initiation
  The quality-adjusted time without symptoms or toxicity (Q-TWiST) integrates data from patient-reported outcomes (PROs) into survival calculations. It quantifies the utility-weighted sum of mean time across three health states: time with all-cause grade 3/4 toxicity prior to progression, time without grade 3/4 toxicity or symptoms of progression, and time after progression.
Cost-effectiveness | 24 months from treatment initiation
  Measured by the incremental cost-effectiveness ratio (ICER) to provide the ratio of incremental cost per additional quality-adjusted life year (QALY).
Distribution of treatment modality after progression | 36 months from treatment initiation
  Proportion of participants receiving surveillance, focal treatment, or systemic therapy after disease progression.
Objective response rate (ORR) after restarting treatment | 6 months after restarting therapy
  Proportion of participants achieving CMR or PMR per PERCIST 1.0 within 6 months of restarting therapy after progression.

OTHER OUTCOMES:
Metabolic response assessed by serial PET/CT | Baseline to 24 months from treatment initiation
  Metabolic response and changes of FDG-uptake values on serial PET/CT during this trial will be assessed and documented.
Biobanking for future research | Baseline to 24 months from treatment initiation
  Collection of serial peripheral blood samples and other biologic specimens during the trial for subsequent exploratory biomarker studies.

CONTACTS AND LOCATIONS:
Overall Officials: Le Qu, Study Chair — Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, China
Locations (1):
- Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, China, Nanjing, Jiangsu, China